CLINICAL TRIAL: NCT03597984
Title: PREST: Pain REduction With Bone Metastases STereotactic Radiotherapy: A Phase III Randomized Multicentric Trial
Brief Title: Reduction of Pain Symptoms With Stereotactic Radiotherapy on Bone Metastases
Acronym: PREST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Dr. Cellini, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0013663/18
Record Dates: First submitted 2018-05-31; First posted 2018-07-24 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Bone Metastases; Radiotherapy; Technology

STUDY DESIGN:
Intervention Model Description: The study is a randomized, controlled superiority trial. The study will appear as an interventionist without medicinal, multicentric, spontaneous. Randomization will take place in a 1: 1 ratio. The study involves the enrollment of 330 patients divided into two groups of 165 patients for each of the two study arms (arm A (gold standard): 4 Gy x 5 fractions (fr); arm B: 5 Gy x 3 fr (Whole Vertebra) + SIB 10 Gy x 3 fr on the Gross Tumor Volume - GTV). The expected difference between the two treatments in terms of three-month pain control rates is 15% more in the experimental arm compared to the standard arm.
  The calculation of the sample size took into account a 95% CI with a coefficient α of 0.05 and a drop-out rate of 10%.
Who Masked: Participant
Masking Description: For each patient the following variables for balancing the study arms will be considered: Gender, age, performance status, histology, site and primary tumor and presence of visceral metastases; Randomization will be performed at the Gemelli ART of the Gemelli Polyclinic Foundation and will be done by e-mail. Patients will be randomized after verification of inclusion and exclusion criteria. Randomization will be performed according to a random list generated by the computer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (No Intervention): Standard Radiotherapy: 4 Gy x 5 fractions (fr) to Whole vertebra
- Arm B (Experimental): Intervention: Radiotherapy with Simultaneous Integrated Boost-SIB on macroscopic metastases
  Delivery of a boost on macroscopic secondary lesion with Simultaneous Integrated Boost technique according this schedule:
  - 5 Gy x 3 fr (Whole Vertebra) + SIB 10 Gy x 3 fr on the macroscopic disease Gross Tumor Volume - (GTV)
  Interventions: Radiation: Simultaneous Integrated Boost-SIB on macroscopic metastases

INTERVENTIONS:
Radiation: Simultaneous Integrated Boost-SIB on macroscopic metastases — Delivery of a boost on macroscopic secondary lesion with Simultaneous Integrated Boost technique according this schedule:
  - 5 Gy x 3 fr (Whole Vertebra) + SIB 10 Gy x 3 fr on the macroscopic disease Gross Tumor Volume - (GTV)
  Arms: Arm B

SUMMARY:
Interventional study without medicinal, randomized 1: 1 open-label, multicenter, phase 3 to evaluate the response in terms of reduction of pain symptomatology from bone metastases, comparing the conformational radiotherapy (3D-CRT) administered in conventional fractionation vs. extracranial stereotactic radiotherapy (SBRT) administered with concomitant integrated simultaneous boost (Simultaneous Integrated Boost-SIB)

DETAILED DESCRIPTION:
Palliative antalgic oncological treatments, e.g. For patients in the chronic-evolutionary phase of the disease with need for pain control, are a serious problem from the point of view: management, clinical and scientific research. However, they are affecting an ever-increasing volume of patients due to the increased incidence of cancer in all its phases and the potential chronicity of illness linked to new therapies.

The use of palliative anti-radiation radiotherapy treatments potentially involves up to 40% of patients in a Radiotherapy Center. Radiotherapy is commonly used in palliative treatment of symptomatic bone metastases (Furfari A, 2017) being an effective treatment to improve symptoms and consequently improve the quality of life (QoL) of these patients. Due to the peculiar characteristics of the patients who need these treatments, scientific research aimed at optimizing these therapies is a need for assistance and even ethics.

Ideally, this treatment should be as short as possible to re-direct them to systemic therapies or to home care or long-term care systems (e.g.: Hospice). In order to deliver a clinically effective dose in a short period of time, hypofractionated regimens must be used. Stereotactic radiotherapy is a type of radiotherapy that allows to deliver a high equivalent biological dose in a highly conformed manner, with a favorable toxicity profile (Correa RJ, 2016), and generally in a few fractions. The possibility of using special techniques such as stereotactic radiotherapy has been investigated in several phase 2 studies, in terms of symptom response with good results at 3 months (van der Velden JM, 2016) (Murai T1, 2014) (Braam P , 2016) (Deodato F, 2014) (Ryu S, 2014). Further studies have suggested, in order to better manage the toxicity profile linked to the hypofractioned regimen, the possibility of using a hypofractionated regimen over the entire bone compartment and going to over-dose with a stereotaxic regimen only the macroscopically visible disease to the instrumental examinations. In particular, in patients with favorable prognostic scores, this regimen would improve the possible onset of acute and late complications. Although there are indications in the literature (generated by the Consensus Conference) about the radiation treatment schedules to be preferred, there is no globally coded and clinically applied therapeutic prescription standard (Chow E1 & Party, 2012). The most commonly applied conventional radiation treatment schedules include: i) 8 Gy in 1 therapy session; ii) 20 Gy in 5 therapy sessions; iii) 30 Gy in 10 therapy sessions.

With the same pain control, multiple fractionation boards report, according to some authors, better symptom control over time and are therefore very often preferred for patients with a prognosis> 6 months. Routine use of prognostic scores to characterize life expectancy and define the most appropriate treatment regimen is very rarely used in everyday clinical practice.

Modern oncology radiotherapy can take advantage of advanced technologies and exploit the personalization of treatments. To date, some randomized trials are underway investigating the role of stereotactic radiotherapy for these patients compared to conventional approaches, but not all of them use adequate personalization of treatment. Furthermore, none of the ongoing and currently registered trials analyzes the "ii) 20 Gy in 5 treatment sessions" versus stereotactic in the direct comparison between two single randomized arms. The aim of this randomized multicenter prospective trial study is to evaluate the pain control effectiveness of an unconventional fractionation delivered with the most innovative stereotactic technique approach available in this clinical scenario against the conventional one; enrollment of patients will be specifically selected with prognosis> 6 months according to the Mizumoto score (Mizumoto M, 2008) and structural stability defined according to Spine Instability Neoplastic Score (SINS) <7, with indication to radiotherapy on bone metastases. Highlights of this study include: the high level of treatment customization for both accurate selection and ultraconformed radiation therapy planning; the reduction in the number of sessions to which the patient must be subjected, which reduces his discomfort; the approach innovation; the location of the study group (multicentric, in the Italian panorama) in a central position in the international scenario of the specific sector. The results of this trial are potentially "practice-changing".

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with spinal bone metastases from solid, uncomplicated tumor
* Established primary or secondary tumor histology related to the treatment lesion
* Patients aged> 18 years
* Obtaining informed consent
* ECOG 0-2
* Symptomatic patients (NRS> = 4) at the treatment site
* Spine Instability Neoplastic Score (SINS) <7
* Prognosis> 6 months according to Mizumoto Prognostic Score (i.e. Class A and B)
* Spinal metastases verified at MRI including the sites to be enrolled
* No more than 3 non-contiguous spinal segments (e.g. separated by at least two metamers) involved in the study

Exclusion Criteria:

* Impossibility to assign specific NRS for each CTV to be enrolled
* Impossibility to express autonomous consent to therapies
* Pregnancy
* Patient in Hospice or with prognosis <6 months
* Unavailability forecast for 3 month follow-up
* Absence of MRI pre-treatment study
* Impossibility to maintain the treatment position for SBRT
* Previous radiotherapy at the same site or at the level of adjoining metamers (higher or lower than the one to be enrolled)
* Radiometabolic therapy
* Previous enrollment of the same patient for 3 irradiated lesions
* Epidural compression of the spinal cord or of the cauda equina
* Injuries affecting> 25% of the medullary canal and / or a distance <5 mm from the medulla or from the cauda
* Injuries with indication of surgical stabilization
* Chemotherapy or target therapy within the previous 7 days and 7 days after SBRT

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-07-01 (Actual); Study Completion 2020-12-28 (Estimated)

PRIMARY OUTCOMES:
Pain control [EFFICACY and PAIN] | 3 months
  Pain control measured with Numeric Rating Scale (NRS) score, a 11-point scale for patient self-reporting of pain.
  NRS score presents a total range between 0 (no pain) and 10 maximum pain.
  NRS subscale are the sequent:
  * 0: no pain [better outcome ]
  * 1-3: mild pain
  * 4-6: moderate pain
  * 7-10 severe pain [worse outcome]

SECONDARY OUTCOMES:
Pain control duration [EFFICACY and PAIN] | 12 months after end of radiotherapy
  Interval from the end of the RT to the relapse of the symptom
Local control [EFFICACY] | At 3, 6 and 12 months from the end of radiotherapy
  Control of local disease with diagnostic exams according to RECIST 1.1 Criteria
Symptom Progression Free Survival (SPFS) [EFFICACY and PAIN] | 12 months after end of radiotherapy
  Interval from the end of radiotherapy and progressive disease with symptoms according to the criteria of Chow et al. in 2012
Progression-free survival - PFS [EFFICACY] | 12 months
  Interval from the end of radiotherapy and new disease progression
Overall survival [EFFICACY] | 12 months
  Interval between the end of radiotherapy and death
Quality of Life (QoL) [EFFICACY and QUALITY OF LIFE] | At first visit, 1 month and 3 months after the end of radiotherapy
  QoL score according to European Organization for Research and Treatment of Cancer (EORTC): QLQ-C15-PAL
Rate of retreatments [EFFICACY] | 12 months after end of radiotherapy
  Interval from the end of the RT to the start of retreatment

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cellini, MD, Principal Investigator — Fondazione Policlinico Gemelli IRCCS - Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Benedict SH, Yenice KM, Followill D, Galvin JM, Hinson W, Kavanagh B, Keall P, Lovelock M, Meeks S, Papiez L, Purdie T, Sadagopan R, Schell MC, Salter B, Schlesinger DJ, Shiu AS, Solberg T, Song DY, Stieber V, Timmerman R, Tome WA, Verellen D, Wang L, Yin FF. Stereotactic body radiation therapy: the report of AAPM Task Group 101. Med Phys. 2010 Aug;37(8):4078-101. doi: 10.1118/1.3438081. PMID 20879569
- [Result] Bentzen SM, Constine LS, Deasy JO, Eisbruch A, Jackson A, Marks LB, Ten Haken RK, Yorke ED. Quantitative Analyses of Normal Tissue Effects in the Clinic (QUANTEC): an introduction to the scientific issues. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S3-9. doi: 10.1016/j.ijrobp.2009.09.040. PMID 20171515
- [Result] Braam P, Lambin P, Bussink J. Stereotactic versus conventional radiotherapy for pain reduction and quality of life in spinal metastases: study protocol for a randomized controlled trial. Trials. 2016 Feb 2;17:61. doi: 10.1186/s13063-016-1178-7. PMID 26829933
- [Result] Chow E, Hoskin P, Mitera G, Zeng L, Lutz S, Roos D, Hahn C, van der Linden Y, Hartsell W, Kumar E; International Bone Metastases Consensus Working Party. Update of the international consensus on palliative radiotherapy endpoints for future clinical trials in bone metastases. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1730-7. doi: 10.1016/j.ijrobp.2011.02.008. Epub 2011 Apr 12. PMID 21489705
- [Result] Correa RJ, Salama JK, Milano MT, Palma DA. Stereotactic Body Radiotherapy for Oligometastasis: Opportunities for Biology to Guide Clinical Management. Cancer J. 2016 Jul-Aug;22(4):247-56. doi: 10.1097/PPO.0000000000000202. PMID 27441744
- [Result] Deodato F, Cilla S, Macchia G, Torre G, Caravatta L, Mariano G, Mignogna S, Ferro M, Mattiucci GC, Balducci M, Frascino V, Piermattei A, Ferrandina G, Valentini V, Morganti AG. Stereotactic radiosurgery (SRS) with volumetric modulated arc therapy (VMAT): interim results of a multi-arm phase I trial (DESTROY-2). Clin Oncol (R Coll Radiol). 2014 Dec;26(12):748-56. doi: 10.1016/j.clon.2014.08.005. Epub 2014 Aug 29. PMID 25175042
- [Result] Furfari A, Wan BA, Ding K, Wong A, Zhu L, Bezjak A, Wong R, Wilson CF, DeAngelis C, Azad A, Chow E, Charames GS. Genetic biomarkers associated with pain flare and dexamethasone response following palliative radiotherapy in patients with painful bone metastases. Ann Palliat Med. 2017 Dec;6(Suppl 2):S240-S247. doi: 10.21037/apm.2017.09.04. Epub 2017 Sep 20. PMID 29156912
- [Result] Guckenberger M, Hawkins M, Flentje M, Sweeney RA. Fractionated radiosurgery for painful spinal metastases: DOSIS - a phase II trial. BMC Cancer. 2012 Nov 19;12:530. doi: 10.1186/1471-2407-12-530. PMID 23164174
- [Result] Mizumoto M, Harada H, Asakura H, Hashimoto T, Furutani K, Hashii H, Takagi T, Katagiri H, Takahashi M, Nishimura T. Prognostic factors and a scoring system for survival after radiotherapy for metastases to the spinal column: a review of 544 patients at Shizuoka Cancer Center Hospital. Cancer. 2008 Nov 15;113(10):2816-22. doi: 10.1002/cncr.23888. PMID 18846565
- [Result] Murai T, Murata R, Manabe Y, Sugie C, Tamura T, Ito H, Miyoshi Y, Shibamoto Y. Intensity modulated stereotactic body radiation therapy for single or multiple vertebral metastases with spinal cord compression. Pract Radiat Oncol. 2014 Nov-Dec;4(6):e231-7. doi: 10.1016/j.prro.2014.02.005. Epub 2014 Mar 31. PMID 25407874
- [Result] Ryu S, Pugh SL, Gerszten PC, Yin FF, Timmerman RD, Hitchcock YJ, Movsas B, Kanner AA, Berk LB, Followill DS, Kachnic LA. RTOG 0631 phase 2/3 study of image guided stereotactic radiosurgery for localized (1-3) spine metastases: phase 2 results. Pract Radiat Oncol. 2014 Mar-Apr;4(2):76-81. doi: 10.1016/j.prro.2013.05.001. Epub 2013 Jun 4. PMID 24890347
- [Result] van der Velden JM, Verkooijen HM, Seravalli E, Hes J, Gerlich AS, Kasperts N, Eppinga WS, Verlaan JJ, van Vulpen M. Comparing conVEntional RadioTherapy with stereotactIC body radiotherapy in patients with spinAL metastases: study protocol for an randomized controlled trial following the cohort multiple randomized controlled trial design. BMC Cancer. 2016 Nov 21;16(1):909. doi: 10.1186/s12885-016-2947-0. PMID 27871280
- [Derived] Cellini F, Manfrida S, Deodato F, Cilla S, Maranzano E, Pergolizzi S, Arcidiacono F, Di Franco R, Pastore F, Muto M, Borzillo V, Donati CM, Siepe G, Parisi S, Salatino A, D'Agostino A, Montesi G, Santacaterina A, Fusco V, Santarelli M, Gambacorta MA, Corvo R, Morganti AG, Masiello V, Muto P, Valentini V. Pain REduction with bone metastases STereotactic radiotherapy (PREST): A phase III randomized multicentric trial. Trials. 2019 Oct 28;20(1):609. doi: 10.1186/s13063-019-3676-x. PMID 31661034